CLINICAL TRIAL: NCT06537882
Title: A Double-blind Randomized Placebo-controlled Study to Evaluate the Effect of Synbiotics SLP07 on Metabolic Dysfunction-Associated Fatty Liver Disease (MAFLD-RCT)
Brief Title: Evaluate the Effect of Synbiotics on MAFLD
Acronym: MAFLD-RCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GenieBiome Limited (Industry)
Collaborators: Microbiota I-Centre (MagIC) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MAFLD-RCT
Record Dates: First submitted 2024-07-29; First posted 2024-08-05 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Metabolic Dysfunction-Associated Fatty Liver Disease
Keywords: Metabolic dysfunction-Associated Fatty Liver Disease; Synbiotics

STUDY DESIGN:
Intervention Model Description: All subjects will be randomized into two groups to take SLP07 or placebo daily for 3 months with monthly assessment.
Who Masked: Participant, Investigator
Masking Description: Attending physicians, investigators performing assessments in clinic visits and study participants will be blinded to the group allocation until study completion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active arm (Active Comparator): Subjects will take 1 sachet of G-NiiB synbiotics formula (SLP07) daily for 3 months
  Interventions: Dietary Supplement: G-NiiB synbiotics formula (SLP07)
- Placebo arm (Placebo Comparator): Subjects will take 1 sachet of active vitamin daily for 3 months
  Interventions: Dietary Supplement: Active placebo

INTERVENTIONS:
Dietary Supplement: G-NiiB synbiotics formula (SLP07) — SLP07 consists of a blend of food-grade Bifidobacterium and Lactobacillus as active probiotics, omega 3, and vitamin E.
  Arms: Active arm
Dietary Supplement: Active placebo — Active placebo contains 2mg of vitamin C with corn starch filler
  Arms: Placebo arm

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is one of the most common chronic liver diseases worldwide. Available data indicates that probiotics may regulate the gut microbiota, while Vitamin E and omega 3 are safe and effective at treating NAFLD patients. In this study, investigators aim to investigate if the enhanced synbiotic preparation of SLP07 is efficacious in liver function improvement in subjects with MAFLD.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is one of the most common chronic liver diseases worldwide.(1) The prevalence of NAFLD is estimated to be about 20%-30% in the Western world (2) and increasing in Asia. The prevalence of NAFLD across Asia varies from 5% to 40%.(3,4) The population prevalence of NAFLD in Hong Kong Chinese was 27.3%.(1) NAFLD may progress to non-alcoholic steatohepatitis (NASH), cirrhosis, liver failure and liver cancer, and is believed to be the leading etiology for cryptogenic cirrhosis.(5,6) NAFLD is also strongly associated with obesity and metabolic syndrome and is shown to be an independent cardiovascular risk factor.(7,8) Recently, a consensus by an international panel of experts recommended a change in name for NAFLD to metabolic dysfunction associated with fatty liver disease (MAFLD).(9) Patients who fulfil the MAFLD criteria have more severe metabolic and liver disease than those who fulfil the NAFLD criteria alone. At present, there is no standard pharmacologic therapy available for NAFLD or MAFLD currently.

Recently, it has been reported that NAFLD might be linked to small intestinal bacterial overgrowth (SIBO), which induces liver injury by gut-derived lipopolysaccharides (LPS) and TNF- α production. (10) Probiotics have several anti-inflammatory effects that can contribute to their clinical benefits in NAFLD.(11) Gut microbiota also plays a role in the development of insulin resistance, hepatic steatosis, necroinflammation and fibrosis. (12) The use of probiotics, prebiotics and synbiotics has been considered a potential and promising strategy to regulate the gut microbiota.(13,14) In the meantime, Vitamin E has been recommended for use in NAFLD treatmentand prevents liver injury. Moreover, many clinical trials and meta-analyses have evaluated the efficacy of omega 3 (C20-22 ω3 polyunsaturated fatty acids (PUFA)) in reducing existing NAFLD in adults and children, and the results indicate that omega 3 is safe and effective at lowering liver fat in NAFLD patients. (15,16)

In this study, investigators aim to investigate if the SLP07, which is an investigational product that contains a blend of naturally occurring food-grade Bifidobacterium and Lactobacillus strains, omega-3 and vitamin E, is efficacious in liver function improvement in subjects with MAFLD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with MAFLD with CAP ≥ 270 by fibroscan
* Age ≥ 50
* Subjects with diabetes or components of metabolic syndrome
* Subjects have been taking stable medication 3 months prior to enrolment and are expected to remain stable throughout the study period
* Written informed consent can be obtained

Exclusion Criteria:

* Known history of any secondary causes of MAFLD including alcoholic liver disease, drug-induced liver injury, autoimmune hepatitis, viral hepatitis, cholestatic liver disease and metabolic/genetic liver disease
* Active malignancy (on any kind of treatments for the known cancer)
* Known diabetes with poor control (HbA1c > 8.5%) within 3 months
* Significant alcohol consumption (over 10g per day: a half pint or half bottle of beer or a standard-size wine glass)
* Subjects who are using insulin and Glucagon-like peptide-1(GLP1) such as dulaglutide, semaglutide
* Consumption of systemic corticosteroids or methotrexate in the last 6 months
* Use of antibiotics, probiotics or prebiotics one month prior to enrolment
* Taking any supplements which are claimed to possibly protect the liver or improve liver functions including vitamin E and omega-3
* Any condition or allergy history for probiotics
* Any allergy to vitamin E, omega-3 or lactose

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2024-05-17 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with a reduction of at least 1 grade of steatosis AND/OR >10% reduction in CAP scores at 3 months | 3 months
  The change of CAP score measured by fibroscan. CAP score is a measurement of fat accumulation in the liver to further determine the steatosis grade. The CAP score ranges from 100 to 400 decibels per meter (dB/m). The higher the score, the more the steatosis is.

SECONDARY OUTCOMES:
Percentage of participants with improvement in steatohepatitis across the study period. | 3 months
  The percentage of improvement in steatohepatitis compared to the baseline
Change in lipid profile across the study period. | 3 months
  The change in the level of lipid profiles
Change of body mass index (BMI) across the study period. | 3 months
  The change of body weight and body height
Change of body waist circumference across the study period. | 3 months
  The change of waist circumference
Adverse events reported during the study period. | 3 months
  The adverse events reported throughout the study
Changes in faecal microbial profiling across 16 weeks | 3 months
  The change of microbial profile in stool compared to baseline
Change of CAP score across the study period | 3 months
  CAP score is a measurement of fat accumulation in the liver to further determine the steatosis grade. The CAP score ranges from 100 to 400 decibels per meter (dB/m). The higher the score, the more the steatosis is.
Change of liver stiffness (measured in kPa) across the study period | 3 months
  The change of liver stiffness (measured in kPa)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Ching, PhD, Study Director — GenieBiome Limited
Locations (1):
- GenieBiome Limited, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wong VW, Chu WC, Wong GL, Chan RS, Chim AM, Ong A, Yeung DK, Yiu KK, Chu SH, Woo J, Chan FK, Chan HL. Prevalence of non-alcoholic fatty liver disease and advanced fibrosis in Hong Kong Chinese: a population study using proton-magnetic resonance spectroscopy and transient elastography. Gut. 2012 Mar;61(3):409-15. doi: 10.1136/gutjnl-2011-300342. Epub 2011 Aug 16. PMID 21846782
- [Background] Bellentani S, Scaglioni F, Marino M, Bedogni G. Epidemiology of non-alcoholic fatty liver disease. Dig Dis. 2010;28(1):155-61. doi: 10.1159/000282080. Epub 2010 May 7. PMID 20460905
- [Background] Amarapurkar DN, Hashimoto E, Lesmana LA, Sollano JD, Chen PJ, Goh KL; Asia-Pacific Working Party on NAFLD. How common is non-alcoholic fatty liver disease in the Asia-Pacific region and are there local differences? J Gastroenterol Hepatol. 2007 Jun;22(6):788-93. doi: 10.1111/j.1440-1746.2007.05042.x. PMID 17565631
- [Background] Chitturi S, Wong VW, Farrell G. Nonalcoholic fatty liver in Asia: Firmly entrenched and rapidly gaining ground. J Gastroenterol Hepatol. 2011 Jan;26 Suppl 1:163-72. doi: 10.1111/j.1440-1746.2010.06548.x. PMID 21199528
- [Background] Caldwell SH, Oelsner DH, Iezzoni JC, Hespenheide EE, Battle EH, Driscoll CJ. Cryptogenic cirrhosis: clinical characterization and risk factors for underlying disease. Hepatology. 1999 Mar;29(3):664-9. doi: 10.1002/hep.510290347. PMID 10051466
- [Background] Farrell GC, Larter CZ. Nonalcoholic fatty liver disease: from steatosis to cirrhosis. Hepatology. 2006 Feb;43(2 Suppl 1):S99-S112. doi: 10.1002/hep.20973. PMID 16447287
- [Background] Hamaguchi M, Kojima T, Takeda N, Nagata C, Takeda J, Sarui H, Kawahito Y, Yoshida N, Suetsugu A, Kato T, Okuda J, Ida K, Yoshikawa T. Nonalcoholic fatty liver disease is a novel predictor of cardiovascular disease. World J Gastroenterol. 2007 Mar 14;13(10):1579-84. doi: 10.3748/wjg.v13.i10.1579. PMID 17461452
- [Background] Wong VW, Wong GL, Yip GW, Lo AO, Limquiaco J, Chu WC, Chim AM, Yu CM, Yu J, Chan FK, Sung JJ, Chan HL. Coronary artery disease and cardiovascular outcomes in patients with non-alcoholic fatty liver disease. Gut. 2011 Dec;60(12):1721-7. doi: 10.1136/gut.2011.242016. Epub 2011 May 20. PMID 21602530
- [Background] Eslam M, Sanyal AJ, George J; International Consensus Panel. MAFLD: A Consensus-Driven Proposed Nomenclature for Metabolic Associated Fatty Liver Disease. Gastroenterology. 2020 May;158(7):1999-2014.e1. doi: 10.1053/j.gastro.2019.11.312. Epub 2020 Feb 8. PMID 32044314
- [Background] Loguercio C, De Simone T, Federico A, Terracciano F, Tuccillo C, Di Chicco M, Carteni M. Gut-liver axis: a new point of attack to treat chronic liver damage? Am J Gastroenterol. 2002 Aug;97(8):2144-6. doi: 10.1111/j.1572-0241.2002.05942.x. No abstract available. PMID 12190198
- [Background] Solga SF, Diehl AM. Non-alcoholic fatty liver disease: lumen-liver interactions and possible role for probiotics. J Hepatol. 2003 May;38(5):681-7. doi: 10.1016/s0168-8278(03)00097-7. No abstract available. PMID 12713883
- [Background] Eslamparast T, Eghtesad S, Hekmatdoost A, Poustchi H. Probiotics and Nonalcoholic Fatty liver Disease. Middle East J Dig Dis. 2013 Jul;5(3):129-36. PMID 24829682
- [Background] Pandey KR, Naik SR, Vakil BV. Probiotics, prebiotics and synbiotics- a review. J Food Sci Technol. 2015 Dec;52(12):7577-87. doi: 10.1007/s13197-015-1921-1. Epub 2015 Jul 22. PMID 26604335
- [Background] Yadav MK, Kumari I, Singh B, Sharma KK, Tiwari SK. Probiotics, prebiotics and synbiotics: Safe options for next-generation therapeutics. Appl Microbiol Biotechnol. 2022 Jan;106(2):505-521. doi: 10.1007/s00253-021-11646-8. Epub 2022 Jan 11. PMID 35015145
- [Background] Jump DB, Lytle KA, Depner CM, Tripathy S. Omega-3 polyunsaturated fatty acids as a treatment strategy for nonalcoholic fatty liver disease. Pharmacol Ther. 2018 Jan;181:108-125. doi: 10.1016/j.pharmthera.2017.07.007. Epub 2017 Jul 16. PMID 28723414
- [Background] Spooner MH, Jump DB. Omega-3 fatty acids and nonalcoholic fatty liver disease in adults and children: where do we stand? Curr Opin Clin Nutr Metab Care. 2019 Mar;22(2):103-110. doi: 10.1097/MCO.0000000000000539. PMID 30601174